CLINICAL TRIAL: NCT01493596
Title: A Phase 1, Double-blind, Placebo-controlled, Single Ascending Dose Study of the Safety, Tolerability and Pharmacokinetics of CPP-115 Solution Administered Orally to Healthy Volunteers
Brief Title: A Safety, Tolerability and Pharmacokinetic Study of CPP-115
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Catalyst Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CPP-115-0001
Record Dates: First submitted 2011-11-28; First posted 2011-12-16 (Estimated); Results first posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Cocaine Dependency
Keywords: Safety; Tolerability
MeSH Terms: interventions — (1S,3S)-3-amino-4-difluoromethylenecyclopentanecarboxylic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- CPP-115 Dose 1 (Other): Each dose cohort will consist of 8 subjects with 6 subjects randomized to receive CPP-115 and 2 subjects to receive matching placebo. Progression to the next higher dose level will be contingent upon demonstration of a satisfactory assessment of the data from the previous dose.
  Interventions: Drug: CPP-115; Drug: Placebo
- CPP-115 Dose 2 (Other): 2 subjects to receive matching placebo. Progression to the next higher dose level will be contingent upon demonstration of a satisfactory assessment of the data from the previous dose.
  Interventions: Drug: CPP-115; Drug: Placebo
- CPP-115 Dose 3 (Other): Each dose cohort will consist of 8 subjects with 6 subjects randomized to receive CPP-115 and 2 subjects to receive matching placebo. Progression to the next higher dose level will be contingent upon demonstration of a satisfactory assessment of the data from the previous dose.
  Interventions: Drug: CPP-115; Drug: Placebo
- CPP-115 Dose 4 (Other): Each dose cohort will consist of 8 subjects with 6 subjects randomized to receive CPP-115 and 2 subjects to receive matching placebo. Progression to the next higher dose level will be contingent upon demonstration of a satisfactory assessment of the data from the previous dose.
  Interventions: Drug: CPP-115; Drug: Placebo
- CPP-115 Dose 5 (Other): Each dose cohort will consist of 8 subjects with 6 subjects randomized to receive CPP-115 and 2 subjects to receive matching placebo. Progression to the next higher dose level will be contingent upon demonstration of a satisfactory assessment of the data from the previous dose.
  Interventions: Drug: CPP-115; Drug: Placebo
- CPP-115 Dose 6 (Other): Each dose cohort will consist of 8 subjects with 6 subjects randomized to receive CPP-115 and 2 subjects to receive matching placebo. Progression to the next higher dose level will be contingent upon demonstration of a satisfactory assessment of the data from the previous dose.
  Interventions: Drug: CPP-115; Drug: Placebo

INTERVENTIONS:
Drug: CPP-115 — Appropriate amount of drug substance will be dissolved in juice within 3 hours of dosing.
Drug: Placebo — An equal volume of water mixed with juice will be administered.
  Other Names: CPP-115

SUMMARY:
Primary Objective:

• To evaluate the safety and tolerability of ascending single oral doses of CPP-115

Secondary Objective:

• To determine the pharmacokinetic profiles of CPP-115 following administration of a ascending single oral doses

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent and comply with study procedures and requirements.
2. Males, age 18 to 65 years.
3. Body Mass Index between 19 and 32 kg/m2.
4. Normal systolic blood pressure (BP [90-140 mmHg]), diastolic BP (50 90 mmHg) and heart rate (HR [resting HR 40-90 beats per minute (bpm)]).
5. Willing and able to abstain from drug, alcohol, and tobacco use during study participation.

Exclusion Criteria:

1. Medical history and/or findings on physical examination indicating the presence of clinically significant illness.
2. Clinically significant abnormalities of vital signs or clinical laboratory results (including hematology, chemistry, and urinalysis).
3. Presence or recent history (within 28 days prior to Screening) of active and clinically significant (as judged by the Investigator) gastrointestinal, renal, cardiovascular, hepatic, metabolic, allergic, dermatologic, hematologic, pulmonary, neurological or psychiatric illness or disorder.
4. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs.
5. Clinically significant ECG abnormalities including QTc ≥ 450 msec.
6. Use of any tobacco-containing or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to Screening.
7. Use of any prescription, illegal, or investigational drug within 28 days prior to Day 1.
8. Use of any over-the-counter (OTC) drug, including vitamins, minerals, dietary/herbal supplements, or grapefruit or grapefruit juice within 14 days prior to Day 1.
9. Use of alcohol, caffeine, or poppy seed-containing foods or beverages within 72 hours prior to Day 1.
10. History of recent (within 6 months) drug or alcohol abuse, as defined in DSM IV (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition).
11. Positive urine drug screen, urine cotinine test, or alcohol breath test at Screening or check-in to the clinical study unit (CSU). Subjects with results believed to be false positives can be allowed to screen while results are retested at a specialized laboratory.
12. Positive serology for the surface antigen of Hepatitis B (HBsAg), Hepatitis C (anti HCV), or human immunodeficiency virus (HIV) antibody screen.
13. Donation of blood or plasma to a blood bank or for a clinical study (except for study screening) within 28 days prior to Day 1.
14. Receipt of blood products within 2 months prior to Screening.
15. Any condition or other reason that, in the opinion of the Investigator, would render the subject unsuitable for the clinical study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mardik Donikyan, DO, Principal Investigator — Clinilabs, Inc.
Locations (1):
- Clinilabs, Inc., New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 1 unit. Groups of 8 normal volunteer male subjects were screened & returned to unit evening before they were to receive their specified dose.
Pre-assignment Details: Overnight fast prior to receiving dose
Groups:
- CPP-115 Dose 1: Cohort 1 consisted of 8 subjects with 6 subjects randomized to receive CPP-115 and 2 subjects receiving matching placebo solution. Progression to the next higher dose level was contingent upon demonstration of a satisfactory assessment of safety based on committee review the safety data obtained from this dose.
  Placebo : 5 ml water mixed with ~250 ml juice was administered.
  CPP-115 : Appropriate amount of drug substance dissolved in 5 ml water will be dissolved in ~250 ml juice within 3 hours of dosing.
- CPP-115 Dose 2: Cohort 2a consisted of 8 subjects with 6 subjects randomized to receive CPP-115 and 2 subjects receiving matching placebo solution. Progression to the next higher dose level was contingent upon demonstration of a satisfactory assessment of safety based on committee review the safety data obtained from this dose.
  Placebo : 5 ml water mixed with ~250 ml juice was administered.
  CPP-115 : Appropriate amount of drug substance dissolved in 5 ml water will be dissolved in ~250 ml juice within 3 hours of dosing.
- CPP-115 Dose 2 (Repeat): Cohort 2(b) consisted of 7 subjects with 5 subjects randomized to receive CPP-115 and 2 subjects receiving matching placebo solution. Progression to the next higher dose level was contingent upon demonstration of a satisfactory assessment of safety based on committee review the safety data obtained from this dose.
  Placebo : 5 ml water mixed with ~250 ml juice was administered.
  CPP-115 : Appropriate amount of drug substance dissolved in 5 ml water will be dissolved in ~250 ml juice within 3 hours of dosing.
- CPP-115 Dose 3: Cohort 3 consisted of 8 subjects with 6 subjects randomized to receive CPP-115 and 2 subjects receiving matching placebo solution. Progression to the next higher dose level was contingent upon demonstration of a satisfactory assessment of safety based on committee review the safety data obtained from this dose.
  Placebo : 5 ml water mixed with ~250 ml juice was administered.
  CPP-115 : Appropriate amount of drug substance dissolved in 5 ml water will be dissolved in ~250 ml juice within 3 hours of dosing.
- CPP-115 Dose 4: Cohort 4 consisted of 8 subjects with 6 subjects randomized to receive CPP-115 and 2 subjects receiving matching placebo solution. Progression to the next higher dose level was contingent upon demonstration of a satisfactory assessment of safety based on committee review the safety data obtained from this dose.
  Placebo : 5 ml water mixed with ~250 ml juice was administered.
  CPP-115 : Appropriate amount of drug substance dissolved in 5 ml water will be dissolved in ~250 ml juice within 3 hours of dosing.
- CPP-115 Dose 5: Cohort 5 consisted of 8 subjects with 6 subjects randomized to receive CPP-115 and 2 subjects receiving matching placebo solution. Progression to the next higher dose level was contingent upon demonstration of a satisfactory assessment of safety based on committee review the safety data obtained from this dose.
  Placebo : 5 ml water mixed with ~250 ml juice was administered.
  CPP-115 : Appropriate amount of drug substance dissolved in 5 ml water will be dissolved in ~250 ml juice within 3 hours of dosing.
- CPP-115 Dose 6: Cohort 1 consisted of 8 subjects with 6 subjects randomized to receive CPP-115 and 2 subjects receiving matching placebo solution. Assessment of safety based on committee review the safety data obtained from this dose.
  Placebo : 5 ml water mixed with ~250 ml juice was administered.
  CPP-115 : Appropriate amount of drug substance dissolved in 5 ml water will be dissolved in ~250 ml juice within 3 hours of dosing.
Period: Overall Study
Arm/Group | CPP-115 Dose 1 | CPP-115 Dose 2 | CPP-115 Dose 2 (Repeat) | CPP-115 Dose 3 | CPP-115 Dose 4 | CPP-115 Dose 5 | CPP-115 Dose 6
Started | 8 | 8 | 7 (Repeat of dose cohort because of incidences of hyperkalemia observed in cohort 2(a).) | 8 | 8 | 8 | 8
Completed | 8 | 8 | 7 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects randomized to drug had plasma and urine levels of drug analyzed to produce pharmacokinetic profiles (e.g. time to maximum concentration (Cmax), half life (t1/2), area under the curve (AUC)
Groups:
- Total: Total of all reporting groups
Arm/Group | CPP-115 Dose 1 | CPP-115 Dose 2 | CPP-115 Dose 2 (Repeat) | CPP-115 Dose 3 | CPP-115 Dose 4 | CPP-115 Dose 5 | CPP-115 Dose 6 | Total
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 41
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (13.01) | 32.6 (5.67) | 35.2 (12.11) | 38.8 (4.83) | 40.8 (9.93) | 38.0 (10.6) | 35.5 (7.5) | 36.8 (9.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 41
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 41

OUTCOME MEASURES:

1. Primary Outcome: Safety of Single Oral Doses
Description: Number of subjects with clinically significant changes in vital signs, ECG abnormalities changes of cardiac rhythm, serious or severe AEs, and/or clinically significant changes in clinical laboratory evaluations.
Time Frame: Days 1-3, 8 & 30
Measure: Number; unit: participants
Groups:
- CPP-115 Dose 1 (5mg); CPP-115 Dose 4 (80mg); CPP-115 Dose 5 (200mg); CPP-115 Dose 6 (500mg): Each dose cohort will consist of 8 subjects with 6 subjects randomized to receive CPP-115 and 2 subjects to receive matching placebo. Progression to the next higher dose level will be contingent upon demonstration of a satisfactory assessment of the data from the previous dose.
  CPP-115: Appropriate amount of drug substance will be dissolved in juice within 3 hours of dosing.
  Placebo: An equal volume of water mixed with juice will be administered. There were no deaths or SAEs
- CPP-115 Dose 2 (13mg): 2 subjects to receive matching placebo. Progression to the next higher dose level will be contingent upon demonstration of a satisfactory assessment of the data from the previous dose.
  CPP-115: Appropriate amount of drug substance will be dissolved in juice within 3 hours of dosing.
  Placebo: An equal volume of water mixed with juice will be administered. There were no deaths or SAEs
- CPP-115 Dose 3 (32mg): Each dose cohort will consist of 8 subjects with 6 subjects randomized to receive CPP-115 and 2 subjects to receive matching placebo. Progression to the next higher dose level will be contingent upon demonstration of a satisfactory assessment of the data from the previous dose.
  There were no deaths or SAEs
  CPP-115: Appropriate amount of drug substance will be dissolved in juice within 3 hours of dosing.
  Placebo: An equal volume of water mixed with juice will be administered.
Arm/Group | CPP-115 Dose 1 (5mg) | CPP-115 Dose 2 (13mg) | CPP-115 Dose 3 (32mg) | CPP-115 Dose 4 (80mg) | CPP-115 Dose 5 (200mg) | CPP-115 Dose 6 (500mg)
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: CPP-115 Dose 1 (5mg) vs CPP-115 Dose 2 (13mg) vs CPP-115 Dose 3 (32mg) vs CPP-115 Dose 4 (80mg) vs CPP-115 Dose 5 (200mg) vs CPP-115 Dose 6 (500mg); Descriptive statistics for evaluation of AEs; Test type: Other — Comparison of event rates across dose groups; percentage = 14.3 — There were a total of 5 non-serious adverse events for an AE rate of 14.3%; Descriptive statistics of adverse events

ADVERSE EVENTS:
Time Frame: 30 days
Description: Solicited and all events were considered treatment related. There were no SAEs.
Groups:
- CPP-115 Dose 1; CPP-115 Dose 4; CPP-115 Dose 5; CPP-115 Dose 6: Each dose cohort will consist of 8 subjects with 6 subjects randomized to receive CPP-115 and 2 subjects to receive matching placebo. Progression to the next higher dose level will be contingent upon demonstration of a satisfactory assessment of the data from the previous dose.
  CPP-115: Appropriate amount of drug substance will be dissolved in juice within 3 hours of dosing.
  Placebo: An equal volume of water mixed with juice will be administered. There were no deaths or SAEs
- CPP-115 Dose 2: 2 subjects to receive matching placebo. Progression to the next higher dose level will be contingent upon demonstration of a satisfactory assessment of the data from the previous dose.
  CPP-115: Appropriate amount of drug substance will be dissolved in juice within 3 hours of dosing.
  Placebo: An equal volume of water mixed with juice will be administered. There were no deaths or SAEs
- CPP-115 Dose 3: Each dose cohort will consist of 8 subjects with 6 subjects randomized to receive CPP-115 and 2 subjects to receive matching placebo. Progression to the next higher dose level will be contingent upon demonstration of a satisfactory assessment of the data from the previous dose.
  There were no deaths or SAEs
  CPP-115: Appropriate amount of drug substance will be dissolved in juice within 3 hours of dosing.
  Placebo: An equal volume of water mixed with juice will be administered.
Arm/Group | CPP-115 Dose 1 | CPP-115 Dose 2 | CPP-115 Dose 3 | CPP-115 Dose 4 | CPP-115 Dose 5 | CPP-115 Dose 6
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 1/5 | 0/6 | 1/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPP-115 Dose 1 (N=6) | CPP-115 Dose 2 (N=6) | CPP-115 Dose 3 (N=5) | CPP-115 Dose 4 (N=6) | CPP-115 Dose 5 (N=6) | CPP-115 Dose 6 (N=6)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood CPK increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days